CLINICAL TRIAL: NCT05772390
Title: Partial Breast Re-irradiation in Women with Locally Recurrent Breast Cancer Previously Treated with Conservative Surgery and Whole Breast Irradiation: a Prospective Phase II Clinical Study
Brief Title: Partial Breast Re-irradiation in Women in Women with Locally Recurrent Breast Cancer Previously Treated with Conservative Surgery and Whole Breast Irradiation
Acronym: PBReI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST174.25
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Recurrent
Keywords: Partial re-irradiation; recurrent breast cancer; conservative surgery
MeSH Terms: conditions — Breast Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Partial breast re-irradiation (Experimental): partial breast re-irradiation in patients with local recurrence of breast cancer, previously treated with breast conservative surgery and whole breast radiotherapy. A total dose of 35 Gy in 10 daily fractions, 5 fractions per week, will be prescribed.
  Interventions: Radiation: Partial breast re-irradiation

INTERVENTIONS:
Radiation: Partial breast re-irradiation — partial breast re-irradiation

SUMMARY:
A prospective study of partial breast re-irradiation in patients with local recurrence of breast cancer

DETAILED DESCRIPTION:
Breast cancer is the leading type of cancer in women worldwide. Although advances in treatment have led to an overall reduction in breast cancer mortality, survivors continue to have an ongoing risk of disease recurrence. For women who experience breast recurrence, mastectomy has historically been the only treatment approach offered. However, it has been associated with negative health outcomes, including reduced quality of life, depression and anxiety, and impaired sexual functioning. As a result, there is increasing interest to identify treatment options that include breast preservation. Breast-conserving surgery followed by re-irradiation with partial breast irradiation has recently been found to be a safe alternative to mastectomy for women who have undergone prior whole breast radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Isolated ipsilateral unifocal breast lesions;
2. Histologically confirmed invasive breast carcinoma or carcinoma in situ;
3. Limited size (< 2 cm) without evidence of skin involvement;
4. Negative histologic margins of resection;
5. Negative axillary lymph nodes;
6. No synchronous distant metastases;
7. Bilateral breast mammogram or MRI within 120 days prior to study entry;
8. For invasive in-breast recurrence, no more than 120 days since whole-body (positron emission tomography) PET-CT scan OR CT scan of the chest, abdomen, and pelvis, and bone scan (if clinically relevant);
9. ≥ 24 months interval between initial breast conserving therapy (surgery and whole breast radiotherapy) and recurrence;
10. Female, aged >18 years;
11. Life expectancy of greater than 12 months;
12. ECOG performance status <2;
13. Female participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 4 months thereafter;
14. Participant is willing and able to give informed consent for participation in the study;

Exclusion Criteria:

1. Regional recurrences (axillary, supraclavicular);
2. Positive histologic margins at resection;
3. Metastatic disease;
4. Previous breast RT performed with IORT, brachytherapy or previous partial breast treatment;
5. Known pathogenic mutation of BRCA1, BRCA2 or TP53 gene;
6. Patients who had chemotherapy within 2 weeks prior to study RT;
7. Participation in another clinical trial with any investigational agents within 30 days prior to study screening;
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements;
9. Significant comorbidity precluding RT for breast cancer (cardiovascular or pulmonary disease, sclerodermia, systemic lupus erythematosus);
10. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years (except for previously treated basal cell carcinoma of the skin and in situ carcinoma of the uterine cervix, endometrium or colon);
11. Inaccessibility for follow-up;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Treatment related toxicity | 12 months
  determine the toxicity of partial breast re-irradiation (PBrI) as rate of grade ≥ 3 treatment-related skin, fibrosis, and breast pain Adverse Events, accordin to Common Terminology Criteria for Adverse Events scale 5.0 (Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE) up to 1 year from completion of radiation treatment

SECONDARY OUTCOMES:
in-breast recurrence in the ipsilateral breast | 5 years
  In-breast recurrence is defined histologic evidence of recurrent carcinoma, invasive or noninvasive (excluding lobular carcinoma in situ), in the ipsilateral breast
Number of patients free from mastectomy over total number of patients | 5 years
  Freedom from mastectomy is calculated from mastectomy failure rates. Failure is a mastectomy of the treated breast performed for any reason
To evaluate distant-metastasis free survival | 5 years
  Distant metastasis-free survival is defined as time from registration to the appearance of a distant metastasis confirmed radiographically and/or pathologically or death from any cause
Overall survival | 5 years
  Overall survival is defined as time from registration to date of death or last follow-up
Patient satisfaction | 5 years
  Patients satisfaction is assessed with the Breast-Q questionnaire (from 0 (worst) to 100 (best). Higher scores reflect a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Simona Cima, Study Chair — IRCCS IRST
Locations (1):
- UO Radioterapia, IRST IRCCS, Meldola, Forlì Cesena, Italy

IPD SHARING:
Plan to Share IPD: No